CLINICAL TRIAL: NCT04920266
Title: Validity of a Smart Cap in Measuring Fluid Intake and a Smart Sweat Patch in Measuring Sweat Rate and Sweat Chloride Concentration During Exercise
Brief Title: Validity of Smart Cap and Smart Sweat Patch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2104
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Fluid Intake in Athletes; Sweating Rate in Athletes; Sweat Chloride Concentration in Athletes
Keywords: sweat; hydration; wearable; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Each subject will serve as his or her own control. We will compare the Test and Reference methods during moderate intensity self-paced training runs, coach-led fitness sessions, and/or group outdoor cycling rides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smart sweat patch for sweat rate and sweat chloride concentration (Experimental): Epidermal microfluidic patch that is a flexible 27 cm2 platform with an adhesive backing that collects sweat through a skin-facing inlet port. Custom software uses the smartphone camera to capture and analyze the microfluidic patch.
  Interventions: Device: Sweat Patch, all subjects- running, fitness, cycling
- Reference sweat patch for sweat rate and sweat electrolytes (Placebo Comparator): Regional absorbent patch technique for sweat rate (gravimetry) and electrolytes (sodium, potassium, chloride) by ion chromatography
  Interventions: Device: Reference sweat patch, all subjects - running, fitness, cycling
- Smart Cap bottle fluid measurement (Experimental): Fluid level sensor integrated into the squeeze bottle cap measures the amount of fluid remaining in the bottle via light reflection
  Interventions: Device: Smart Cap, running and fitness exercisers only
- Reference method bottle fluid measurement (Other): Scale weight of bottle (gravimetry method) for Smart Cap bottles (running and fitness subjects) and non-Smart Cap bottles (cyclists)
  Interventions: Other: Bottle Scale, all subjects - running, fitness, cycling

INTERVENTIONS:
Device: Smart Cap, running and fitness exercisers only — Bottle cap
  Arms: Smart Cap bottle fluid measurement
Device: Sweat Patch, all subjects- running, fitness, cycling — Regional contralateral forearm patch
  Arms: Smart sweat patch for sweat rate and sweat chloride concentration
Device: Reference sweat patch, all subjects - running, fitness, cycling — Regional contralateral forearm patch
  Arms: Reference sweat patch for sweat rate and sweat electrolytes
Other: Bottle Scale, all subjects - running, fitness, cycling — Bottle weight
  Arms: Reference method bottle fluid measurement

SUMMARY:
The main objectives are to determine the validity of a Smart Cap in measuring fluid intake during running and fitness exercise and the validity of a Smart Sweat Patch in measuring sweat rate and sweat chloride concentration during outdoor cycling, running, and fitness exercise. A secondary objective is to compare regional sweating rate and sweat electrolyte concentrations (sodium, chloride, and potassium) on contralateral arms with vs. without tattoos.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* Subject is 16-65 years of age
* Subject is moderately-trained (participates in regular outdoor fitness (~1 h), cycling (1-2 h), or running (0.5-1 h) sessions ≥2x per week)
* Subject is participating in an instructor-led fitness session, typical training run, or group bicycle ride

Exclusion Criteria:

* Subject is pregnant
* Subject is a smoker
* Subject is taking a medication or oral supplement that could interfere with study results
* Subject has an allergy to adhesives (e.g., experiences rash reactions to typical adhesive bandages)
* Subject has ≥ 2 cardiovascular risk factors as assessed on the General Health History Questionnaire
* Subject has participated in a clinical trial within past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk
* Subject is employed by, or has a parent, guardian or other immediate family member employed by, a company that manufactures any products that compete with any Gatorade products. If subject is unsure if a company would be considered a competitor to Gatorade they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Fluid intake | Change from baseline to up to 1 hour of exercise
  Smart Cap (sensor) versus Reference method (bottle weight)
Regional sweating rate | Change from baseline to up to 2 hours of exercise
  Sweat Patch versus Reference patch method
Regional sweat chloride concentration | Change from baseline to up to 2 hours of exercise
  Sweat Patch versus Reference patch method

SECONDARY OUTCOMES:
Regional sweating rate with versus without tattoos | Change from baseline to up to 2 hours of exercise
  Reference sweat patch method
Regional sweat sodium and potassium with versus without tattoos | Change from baseline to up to 2 hours of exercise
  Reference sweat patch method
Whole body sweat rate | Body mass change from baseline to up to 2 hours of exercise
  Scale weight

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Principal Investigator — PepsiCo Global R&D, Gatorade Sports Science Institute (GSSI)
Locations (3):
- United States (3):
  - Gatorade Sports Science Institute (GSSI), 617 West Main Street, Barrington, Illinois
  - Grant Park, 337 E Randolph St, Chicago, Illinois
  - Cuba Marsh Forest Preserve, 24205 Cuba Rd, Deer Park, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merritt JR, Ozga M, De Chavez PJD, Boolani A, Baker LB. No effect of tattoos on local sweat concentrations of select cytokines, cortisol, glucose, blood urea nitrogen, or lactate during exercise. Sci Rep. 2024 May 31;14(1):12570. doi: 10.1038/s41598-024-63057-0. PMID 38821996
- [Derived] Keyes DM, Brown SD, King MA, Engel MD, Ciciora-Gold M, Chavez PJD, Baker LB. Multiple regression analyses to determine the effect of sweating rate and tattoo characteristics on sweat outcome measures during exercise. Eur J Appl Physiol. 2022 Oct;122(10):2163-2174. doi: 10.1007/s00421-022-04989-1. Epub 2022 Jul 1. PMID 35778519